CLINICAL TRIAL: NCT06988215
Title: The Effects of Kinesiology Taping Combined With Swallowing Exercises on Oropharyngeal Muscle Thickness and Swallowing Function in Dysphagia Rehabilitation of Stroke Patients: An Ultrasonographic Assessment in a Single-Blind Randomized Controlled Trial
Brief Title: Effect of Kinesiology Taping and Swallowing Exercises on Suprahyoid Muscle Thickness and Swallowing Function in Stroke Patients With Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, elifbusrademirel, Medical Doctor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/26; 2025/26 (Other: Istanbul University-Cerrahpasa Clinical Research Ethics Committee)
Record Dates: First submitted 2025-05-17; First posted 2025-05-23 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Dysphagia; Cerebrovascular Disorders
Keywords: Kinesiology Taping; Dysphagia Rehabilitation; Suprahyoid Muscles; Ultrasound Assessment; Neurogenic Dysphagia
MeSH Terms: conditions — Stroke; Deglutition Disorders; Cerebrovascular Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. The intervention group will receive kinesiology taping combined with swallowing exercises, while the control group will receive placebo taping with the same exercises. Both groups will undergo the intervention for 6 weeks.
Who Masked: Participant
Masking Description: This is a single-blind study in which only the participants are unaware of their group assignment. Participants in both the intervention and control groups receive kinesiology taping; however, only the intervention group receives therapeutic taping while the control group receives placebo taping that appears identical. Care providers and investigators are not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiology Taping Group (Experimental): Participants in this group will receive real kinesiology taping applied to the suprahyoid region along with standardized effortful swallowing and oromotor exercises. The taping will be applied in three directions (hyoid to clavicle, hyoid to sternum, and horizontal to hyoid) and renewed every three days over a 6-week period. Exercises will be performed daily, 5 sets of 10 swallows (50 total repetitions).
  Interventions: Other: Kinesiology Taping with Exercise
- Placebo Taping Group (Placebo Comparator): Participants in this group will receive placebo kinesiology taping that mimics the appearance of therapeutic taping, without applying actual tension. The same standardized swallowing and oromotor exercises will be provided daily for 6 weeks, identical to the experimental group.
  Interventions: Other: Placebo Taping with Exercise

INTERVENTIONS:
Other: Kinesiology Taping with Exercise — Real kinesiology taping is applied to the suprahyoid region in three directions (from the hyoid bone to the clavicle, to the sternum, and horizontally). Taping is renewed every three days. Participants also perform effortful swallowing and oromotor exercises daily (5 sets of 10 repetitions) for 6 weeks.
  Arms: Kinesiology Taping Group
Other: Placebo Taping with Exercise — Non-therapeutic kinesiology taping with no tension is applied to the suprahyoid region to mimic the appearance of the therapeutic tape. Participants perform the same daily swallowing and oromotor exercises as the intervention group for 6 weeks
  Arms: Placebo Taping Group

SUMMARY:
This randomized controlled single-blind study aims to investigate the effect of kinesiology taping combined with resistance exercises on suprahyoid muscle thickness and swallowing function in patients with stroke-related dysphagia. A total of 36 participants will be randomly assigned to an intervention group receiving real kinesiology taping and a control group receiving placebo taping, both combined with standardized swallowing exercises for 6 weeks. Outcome measures include ultrasonographic evaluation of oropharyngeal muscles (geniohyoid, mylohyoid, anterior digastric, and tongue muscles), swallowing function assessed by the Volume-Viscosity Swallow Test, EAT-10, T-SWAL-QOL, Dysphagia Handicap Index, FOIS, and Functional Ambulation Level. This study will contribute to determining effective rehabilitation methods for improving safe swallowing in post-stroke patients.

DETAILED DESCRIPTION:
Dysphagia is a common complication following stroke, associated with serious consequences such as dehydration, malnutrition, and aspiration pneumonia. These complications can prolong hospital stays, impair physical function, and reduce the overall quality of life. The suprahyoid muscle group, which plays a crucial role in the pharyngeal phase of swallowing, is often affected post-stroke. Weakness in these muscles can lead to impaired hyolaryngeal excursion, resulting in incomplete upper esophageal sphincter (UES) opening, residue in the valleculae and piriform sinuses, and increased risk of aspiration and penetration.

The suprahyoid muscles (geniohyoid, mylohyoid, anterior belly of digastric, and stylohyoid) are essential for the anterior-superior movement of the hyolaryngeal complex during swallowing. Rehabilitation targeting this muscle group is clinically important to restore safe and effective swallowing function.

Kinesiology taping (KT) is a non-invasive method widely used in musculoskeletal rehabilitation. KT is believed to support joint alignment, enhance muscle function, and provide mechanical feedback through skin tension. In recent studies, KT has shown promise in enhancing the effects of rehabilitation in conditions such as ankle instability, adhesive capsulitis, and hallux valgus. KT has also been proposed as a novel therapeutic option in the management of neurogenic dysphagia by providing resistance to the hyolaryngeal complex, thereby increasing muscle engagement during swallowing exercises.

This single-blind randomized controlled trial aims to investigate the effects of resistance exercises combined with kinesiology taping on the suprahyoid muscle group in patients with stroke. A total of 36 patients will be randomly assigned into two equal groups: the control group (receiving placebo kinesiology taping plus standard exercises) and the intervention group (receiving real kinesiology taping plus standard exercises).

Ultrasonographic assessment of the suprahyoid muscles (geniohyoid, mylohyoid, anterior digastric, and tongue muscles) will be conducted at baseline and after 6 weeks. Swallowing function will be evaluated using the Volume-Viscosity Swallow Test (VVST), the Eating Assessment Tool (EAT-10), Turkish version of the Swallowing Quality of Life Questionnaire (T-SWAL-QOL), the Dysphagia Handicap Index (DHI), the Functional Oral Intake Scale (FOIS), and the Functional Ambulation Measure (FIM).

Kinesiology tape will be applied in three directions: from the hyoid bone to the clavicle, to the sternum, and horizontally across the hyoid. Participants in both groups will perform effortful swallow and oromotor exercises daily (50 swallows per day, divided into 5 sets of 10 repetitions) for 6 weeks. Tape will be renewed every 3 days.

This study will help determine whether kinesiology taping can enhance the outcomes of dysphagia rehabilitation in post-stroke patients, potentially offering a low-cost and non-invasive adjunctive treatment to traditional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 50 and 80 years
* Diagnosed with stroke
* Mini-Mental State Examination (MMSE) score greater than 22
* Voluntary participation with written informed consent

Exclusion Criteria:

* Open wounds or unresolved skin problems in the neck area
* Known allergy to kinesiology tape or its components
* Medically unstable conditions
* Primary esophageal disorders (e.g., achalasia, upper esophageal sphincter dysfunction)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Measurement of Oropharyngeal Muscle Thickness Time Frame: Baseline and Week 6 Outcome Description: The thickness of oropharyngeal muscles, including the mylohyoid, geniohyoid, anterior belly of digastric, and tongue muscles, will be measured | Baseline and Week 6
  The thickness of oropharyngeal muscles, including the mylohyoid, geniohyoid, anterior belly of digastric, and tongue muscles, will be measured using ultrasonography at baseline and after 6 weeks of intervention.

SECONDARY OUTCOMES:
Change in Swallowing Safety Assessed by Volume-Viscosity Swallow Test (VVST) | Baseline and Week 6
  Swallowing function will be evaluated using the Volume-Viscosity Swallow Test to assess changes in safety and efficiency of oral intake before and after the intervention.
9Change in Dysphagia Severity Assessed by EAT-10(The Eating Assessment Tool | Baseline and Week 6
  The Eating Assessment Tool (EAT-10) will be used to quantify self-perceived dysphagia symptoms. Scores will be compared between baseline and the sixth week.
Change in Swallowing-Related Quality of Life (T-SWAL-QOL) | Baseline and Week 6
  Swallowing-related quality of life will be assessed using the Turkish version of the SWAL-QOL questionnaire, administered before and after the intervention.
Change in Dysphagia Handicap Index (DHI) | Baseline and Week 6
  The Dysphagia Handicap Index will be used to evaluate the psychosocial and functional impact of dysphagia on patients, assessed pre- and post-treatment.
Change in Functional Independence Measure (FIM) | Baseline and Week 6
  The Functional Independence Measure will be used to assess changes in overall functional status and mobility in relation to swallowing performance over the 6-week period.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Büşra Demirel, MD, Principal Investigator — SBÜ Istanbul Physical Medicine and Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training Research Hospital, Istanbul, bahçelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not been finalized. Ethical approval and institutional policies will be reviewed before making a final determination.